CLINICAL TRIAL: NCT03223207
Title: CareLink Express (CLE Research)
Acronym: CLE
Status: Completed | Type: Observational
Sponsor: Baylor Research Institute (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: 015-234
Record Dates: First submitted 2016-02-25; First posted 2017-07-21 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2017-07

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Control Group: The control group will include CIED patients who have been evaluated in the ED at The Heart Hospital Baylor Plano and Baylor Regional Medical Center at Plano. A minimum of 50 devices not compatible with the CareLink Express® system will be prospectively interrogated in the traditional evaluation method using the device manufacturer representative.
- CareLink Express: The study group will include CIED patients who present to the ED and receive a device evaluation using the CareLink Express® system. A minimum of 50 devices will be prospectively evaluated using CareLink Express®.

SUMMARY:
The primary objective of this research is to determine if evaluating CIEDs using CareLink Express® can lead to shorter time to interrogation in the Emergency Department compared to evaluation of devices using traditional evaluation procedures. The goal of the research is to determine if patients evaluated by CareLink Express® have a reduction of "time to interrogation" compared to the traditional patient cohort.

Secondary objectives of the study are to determine any significant differences in the two populations regarding:

1. Health care resource utilization including total charges for ED care.
2. Number of patients leaving the ED without being seen (LWBS) or left without the device interrogation completed.
3. Device related issues detected.

DETAILED DESCRIPTION:
Background:

Over the past 15 years the number of Cardiac Implantable Electronic Devices (CIEDs) implanted has increased dramatically. This is due in part to the aging of the population in general, but primarily due to expanded indications for implantable cardioverter-defibrillators (ICDs), cardiac resynchronization pacemaker therapy (CRT-P) devices, and CRT devices with defibrillator capabilities ("biventricular ICDs" or CRT-D devices). As more patients with structural heart disease survive longer, and as more CIEDs are placed, the number of patients requiring treatment in the emergency departments for arrhythmias and potential device-related matters has increased.

When a patient with a CIED experiences a problem they presume to be cardiac in nature, they often go to the emergency room to seek care. Most emergency departments (ED) are neither equipped to interrogate the CIED, nor staffed with personnel trained to interrogate the CIED. These CIEDs often record data that can assist the physician in the formulation of a diagnostic and treatment strategy tailored to the specific needs of the patient. However, interrogation of the device is dependent on proprietary programming equipment that is not routinely kept in the emergency department. The programming equipment has traditionally been a "stand-alone" unit, which can store the data from the device interrogation (onto a USB drive or floppy disk), but does not have the capability to transmit the data to the patient's physician for rapid interpretation. In addition, ED personnel are not routinely trained to assess CIEDs. In most health care institutions, it is standard practice for a representative of the manufacturer to be contacted so the device can be evaluated. The representative must then travel to the ED with the programming equipment to interrogate the CIED on site. After interrogation, either the representative discusses the findings with the ED physician, or calls the physician that manages the patient's device. The process of in-person device evaluation can be cumbersome and inefficient, especially in an emergency setting. The time involved in the device interrogation process can cause delays in patient care and add unnecessary costs for the patient and health care institution.

Methods:

Patients with CIEDs will be evaluated in the ED setting. Patients will be divided into two cohorts. Each cohort will have a minimum of 50 patients.

The control group will include CIED patients who have been evaluated in the ED at The Heart Hospital Baylor Plano and Baylor Regional Medical Center at Plano. A minimum of 50 devices not compatible with the CareLink Express® system will be prospectively interrogated in the traditional evaluation method using the device manufacturer representative.

The study group will include CIED patients who present to the ED and receive a device evaluation using the CareLink Express® system. A minimum of 50 devices will be prospectively evaluated using CareLink Express®.

The patient's presenting symptoms in the ED include any medical conditions (not just cardiac).

Consent will be obtained from the subject after treatment has occurred in the ED and prior to release. Consent can be obtained from the subject or the subject's Legally Authorized Representative. This will ensure that treatment is not delayed or altered for research purposes.

Initial data will be collected using a Data Collection Form. The research staff or a research trained Emergency Department staff member will complete the Data Form.

Data will be collected by the research coordinators who will collect the Data Collection Forms from the ED at The Heart Hospital Baylor Plano and Baylor Regional Medical Center at Plano. The Data Collection Form will be used by the research coordinators to determine the patient's study cohort.

Other data will be collected by the research coordinators using the hospital EMR and Financial systems.

Data Collection:

Criteria for the hospital and ED encounters will be extracted from the hospital EMR, the Data Collection Form, or the hospital financial system. Device data will be extracted from the device report completed at the time of the device interrogation.

ELIGIBILITY:
Inclusion Criteria:

1) Patients who present to the ED with a problem they believe to be cardiac in nature.

Exclusion Criteria:

1. Patients who present to the ED after transmitting a remote device evaluation within the last 24 hours.
2. Patients referred to the ED from a physician's office or other health care facility where the CIED has already been interrogated or evaluated.
3. Patients in cardiac arrest or other life threatening situations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who arrive to the Emergency Department with a problem they presume to be cardiac in nature.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-08-27 (Actual); Study Completion 2018-08-27 (Actual)

PRIMARY OUTCOMES:
Patients evaluated by CareLink Express have a reduction of "time of interrogation" compared to the traditional patient cohort. | 1 year
  The primary objective of this research is to determine if evaluating CIEDs using CareLink Express® can lead to shorter time to interrogation in the Emergency Department compared to evaluation of devices using traditional evaluation procedures.

SECONDARY OUTCOMES:
Significant differences between the two populations from data analysis | 2 years
  Health care resource utilization including total charges for ED care, number of patients leaving the ED without being seen (LWBS) or left without the device interrogation completed, or device related issues detected.